CLINICAL TRIAL: NCT03027375
Title: Evaluating the Safety and Efficacy of Qishen Granules Among Patients With Chronic Heart Failure: Study Protocol for a Randomized Controlled Trial
Brief Title: Evaluating the Safety and Efficacy of Qishen Granules Among Patients With Chronic Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: China-Japan Friendship Hospital (Other); Zhengzhou Hospital of Traditional Chinese Medicine (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Wei Wang, Vice-President, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-ZXFZJJ-003
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure; Cardiovascular Diseases
Keywords: chronic heart failure; traditional Chinese medicine; Qishen granules
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — qishen granule

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qishen granules (Experimental): The QSG treatment group will receive Qishen granules (13.6 g/pouch, twice per day-30 minutes after breakfast and dinner-for 12 weeks; dosage based on the requirements of Pharmacopoeia of the People's Republic of China).
  Interventions: Drug: Qishen Granules
- placebo granules (Placebo Comparator): The placebo group will receive placebo granules (13.6 g/pouch, twice per day-30 minutes after breakfast and dinner-for 12 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qishen Granules — The QSG are manufactured by Beijing tcmages Pharmaceutical Co., Ltd. (Beijing, China), a company that has obtained Chinese Good Manufacturing Practice for Pharmaceutical Products certification. All the ingredients have been approved by the Chinese Ministry of Food and Drug Safety. 13.6 grams (dry weight) of granules consist of six herbs: Astragalus membranaceus (Fisch.) Bge. var. Mongolicus (Bge.) Hsiao (6g), Salvia miltiorrhiza Bge. (1.5g), Lonicera japonica Thunb. (2g), Scrophularia ningpoensis Hemsl. (2g), Aconitum carmichaeli Debx. (0.9g), and Glycyrrhiza uralensis Fisch. (1.2g).
  Other Names: Yixin Jiedu formula
  Arms: Qishen granules
Drug: Placebo — The placebo is manufactured by Beijing tcmages Pharmaceutical Co., Ltd. (Beijing, China) as well, following the Specification for processing Chinese medicine in Beijing. The placebo granules are similar in appearance, taste, and scent to the Qishen granules.
  Arms: placebo granules

SUMMARY:
This trial will assess the efficacy and safety of QSG in CHF.

DETAILED DESCRIPTION:
Background: Chronic heart failure(CHF), the final stage of various cardiovascular diseases, is a major public health problem associated with significant hospitalization rates, mortality, and huge health care costs, despite advances in the treatment and management of heart failure and heart failure related risk factors. Qishen granules(QSG), a Chinese herbal formula, is widely used by traditional chinese medicine(TCM) practitioners to treat CHF. Several animal experimental studies have showed that QSG can significantly relieve the heart failure symptoms of CHF rat models. However, there is yet no standard clinical trial to assess that. Thus, the investigators are conducting this study to evaluate the efficacy and safety of QSG in a large, varied population.

Methods/Design: This study is designed as a randomized, multi-center, placebo-controlled, double-blind , parallel-group clinical trial. An established total of 200 patients with CHF will be recruited and randomly allocated to either the QSG treatment group or the placebo group (a 1:1 ratio). The patients will receive QSG or placebo granules twice daily for 12 weeks. The primary endpoint is the reduction or percent change in the plasma N-terminal pro-B-type natriuretic peptide(NT-proBNP) level during 12 weeks of treatment. The secondary endpoints consist of composite cardiac events (CCEs), New York Heart Association (NYHA) functional classification, 6-minute walking distance (6MWD), Left ventricular ejection fraction, patient quality of life and TCM syndrome integral scale.

Discussion: This trial will assess the efficacy and safety of QSG in CHF.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years;
2. clinical findings of CHF for at least 3 months prior to screening;
3. CHF caused by coronary heart disease and hypertension, which is diagnosed according to the Chinese guidelines published in 2014 for the diagnosis and management of CHF;
4. clinically stable condition with an NYHA functional class of II to III and an optimal medical treatment with a fixed dosage for at least 2 weeks;
5. a documented left ventricular ejection fraction (LVEF) ≤40% and a serum NT-proBNP level ≥450 pg/ml;
6. CHF of Qi deficiency and blood stasis syndrome;
7. provision of written informed consent.

Exclusion Criteria:

1. CHF complicated with severe valvular disease, congenital heart disease, pericardial disease, cardiomyopathy, unstable angina, acute myocardial infarction(in recent 4 weeks), cardiogenic shock, acute myocarditis, infective endocarditis, uncontrolled severe cardiac arrhythmia with hemodynamic changes;
2. pulmonary heart disease, pulmonary hypertension caused by acute or chronic pulmonary embolism or cerebral apoplexy in recent 6 months;
3. severe hepatic inadequacy with alanine aminotransferase or alkaline phosphatase levels >2 times the upper normal limit, renal inadequacy with a creatinine clearance rate>20% or a serum creatinine level>3mg/dl (>265μmol/L), severe electrolyte imbalance, severe hematologic disease, malignant tumor, diabetes mellitus with severe complications, or severe endocrine diseases such as hyperthyroidism and hypothyroidism;
4. acute infection confirmed by any one of the following 3 tips: 1) fever; 2) a white blood cell count>10×109/L and a percentage of neutrophils>85%; 3) shadows on chest X-ray;
5. uncontrolled blood pressure or fibrosis in other organs;
6. CHF of yin deficiency according to TCM syndrome differentiation;
7. pregnancy or breastfeeding;
8. psychiatric or infectious disease;
9. patients who have participated in other clinical trials in the past two months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the reduction or percent change in the plasma N-terminal pro-B-type natriuretic peptide | 12weeks

SECONDARY OUTCOMES:
composite cardiac events | 4weeks,8weeks,12weeks
New York Heart Association (NYHA) functional classification | 4weeks,8weeks,12weeks
6-minute walking distance | 4weeks,8weeks,12weeks
Left ventricular ejection fraction | 12weeks
Chronic Heart Failure Quality of Life Scale of Integrated Chinese and Western Medicine | 4weeks,8weeks,12weeks
TCM syndrome integral scale | 4weeks,8weeks,12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Study Chair — Beijing University of Chinese Medicine; Huihui Zhao, Doctor, Study Director — Beijing University of Chinese Medicine; Jinping Wang, Master, Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Zhang J, Huang J, Ma A, Yang J, Li W, Wu Z, Yao C, Zhang Y, Yao W, Zhang B, Gao R; Efficacy and Safety of Qili Qiangxin Capsules for Chronic Heart Failure Study Group. A multicenter, randomized, double-blind, parallel-group, placebo-controlled study of the effects of qili qiangxin capsules in patients with chronic heart failure. J Am Coll Cardiol. 2013 Sep 17;62(12):1065-1072. doi: 10.1016/j.jacc.2013.05.035. Epub 2013 Jun 7. PMID 23747768
- [Background] General Assembly of the World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. J Am Coll Dent. 2014 Summer;81(3):14-8. PMID 25951678
- [Background] Switula D. Principles of good clinical practice (GCP) in clinical research. Sci Eng Ethics. 2000 Jan;6(1):71-7. doi: 10.1007/s11948-000-0025-z. PMID 11273440
- [Result] van Riet EE, Hoes AW, Wagenaar KP, Limburg A, Landman MA, Rutten FH. Epidemiology of heart failure: the prevalence of heart failure and ventricular dysfunction in older adults over time. A systematic review. Eur J Heart Fail. 2016 Mar;18(3):242-52. doi: 10.1002/ejhf.483. Epub 2016 Jan 4. PMID 26727047
- [Derived] Du K, Liu J, Tan N, Huang X, Wang J, Zhao H, Wang W. The effects of qishen granules for patients with chronic heart failure: A multicenter randomized double-blind placebo-controlled trial. Front Pharmacol. 2022 Dec 23;13:1017734. doi: 10.3389/fphar.2022.1017734. eCollection 2022. PMID 36618925
- [Derived] Wang J, Shi J, Wei J, Wang J, Gao K, Li X, Chen J, Li S, Zhao H, Wang W. Safety and efficacy of Qishen granules in patients with chronic heart failure: study protocol for a randomized controlled trial. Trials. 2017 Oct 10;18(1):468. doi: 10.1186/s13063-017-2193-z. PMID 29017565